CLINICAL TRIAL: NCT00078741
Title: CBT for PTSD and SMI in Community Mental Health Centers
Brief Title: Cognitive Behavioral Therapy for Post-Traumatic Stress Disorder in Individuals With Severe Mental Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH065248 (NIH); R21MH065248 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2004-03-05; First posted 2004-03-08 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2007-12

CONDITIONS: Stress Disorders, Post-Traumatic; Schizophrenia
Keywords: Psychotic Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Schizophrenia; Psychotic Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT)

SUMMARY:
This study will develop a cognitive behavioral therapy (CBT) program to treat symptoms of post-traumatic stress disorder (PTSD) in people with severe mental illnesses who are treated within community mental health systems.

DETAILED DESCRIPTION:
A significant proportion of people with SMI who are treated within the public sector also suffer from PTSD. Evidence suggests that these individuals often receive inadequate mental health services because effective treatments have not been explored. This study will develop and implement a CBT treatment that is designed specifically for the SMI/PTSD population.

In the first year of the study, a treatment manual and a CBT treatment model, including education, social skills training, and exposure therapy, will be developed. In the following two years, the treatment program will be tested in individuals with SMI and PTSD. Scale ratings, self-report checklists, and daily logs of behavior will be used to assess PTSD symptoms. Scale ratings and self-report surveys will also be used to measure hostility, functional status, depression and schizophrenia symptoms, and satisfaction with the study. Assessments will be made throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD and schizophrenia or schizoaffective disorder
* Active involvement in case management

Exclusion Criteria:

* Suicide risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Frueh, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Department of Mental Health, Columbia, South Carolina